CLINICAL TRIAL: NCT01512355
Title: The Effect of Dexmedetomidine on Decreasing Emergence Agitation and Delirium in Pediatric Patients Undergoing Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2011-0466
Record Dates: First submitted 2012-01-09; First posted 2012-01-19 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Strabismus
MeSH Terms: conditions — Strabismus | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- placebo (Placebo Comparator)
  Interventions: Drug: placebo group

INTERVENTIONS:
Drug: Dexmedetomidine — After, induction of general anesthesia, dexmedetomidine 0.2 mcg/kg/hr continuous intravenous infused during the surgery
  Arms: dexmedetomidine
Drug: placebo group — normal saline_02mcg/kg/hr
  Arms: placebo

SUMMARY:
Postoperative agitation in children is a well-documented clinical phenomenon with incidence ranging from 10% to 67%. Recently, dexmedetomidine has been investigated extensively in the pediatric population and there is now increasing evidence to support the use of this drug as sedative and anesthetic adjunct in children. The purpose of this study is to determine whether prophylactic use of intraoperative dexmedetomidine to prevent of emergence delirium.

ELIGIBILITY:
Inclusion Criteria:

* the patient undergoing the strabismus surgery in severance hospital

Exclusion Criteria:

* delayed development
* mental retardation
* cerebral palsy
* preoperative EKG abnormality e.g. cardiovascular conduction disorder

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
objective pain score | immediate postoperative period up to 1hour after surgery
  1. Objective pain score(OPS) Blood pressure 0~2 points crying 0~2points movement 0~2points agitation 0~2points posture 0~2points complain of pain(where appropiraate by age) 0~2points total 0~10 points
pediatric anesthesia emergence delirium (PAED) scale | immediate postoperative period up to 1hour after surgery
  2. pediatric anesthesia emergence delirium (PAED) scale The Child makes eye contact with the caregiver 0~4 The child's actions are purposeful. 0~4 The child is aware of his'her surroundings. 0~4 The child is restless. 0~4 The child is insonsolable. 0~4 total 0~20 points
5-point agitation scale | immediate postoperative period up to 1hour after surgery
  3. Scoring system for emergence agitation (behavior score)
  1. Sleeping
  2. Awake and calm
  3. Irritable and crying
  4. Inconsolable crying
  5. Severe restlessness and disorientation

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea